CLINICAL TRIAL: NCT01298154
Title: The Effects of Intact and Hydrolyzed Yellow Pea Protein on Food Intake, Glycemic Response, and Subjective Appetite in Healthy Young Men.
Brief Title: Effects of Intact and Hydrolyzed Pea Protein on Food Intake, Glycemic Response and Subjective Appetite
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Dr. Bohdan Luhovyy, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PureNet_23878; peaprotein_486233 (Other Grant/Funding Number: Agriculture & Agri-Food Canada)
Record Dates: First submitted 2010-04-14; First posted 2011-02-17 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Prevention; Obesity Prevention
Keywords: Food intake; Blood glucose; Pulses; Protein
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Intact Pea Protein (20 g) (Experimental)
  Interventions: Other: Dietary intervention
- Hydrolyzed Pea Protein (20 g) (Experimental)
  Interventions: Other: Dietary intervention
- Intact Whey Protein (Experimental)
  Interventions: Other: Dietary intervention
- Hydrolyzed Whey Protein (Experimental)
  Interventions: Other: Dietary intervention
- Water (Experimental)
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Dietary treatments with beverages

SUMMARY:
The purpose of this protocol is to study the effects of intact and hydrolyzed yellow pea protein, compared to intact and hydrolyzed whey protein, on satiety, food intake, and glucose metabolism in healthy young men. The specific objective is to investigate the effects of 20 g available protein for 4 different protein types (intact and hydrolyzed pea and whey proteins) and water (control) on satiety, food intake and blood glucose before and after a meal. The specified amount of protein was chosen based on our previous studies on intact pea protein suggesting that 20 g may reduce food intake and pre-meal blood glucose 30 minutes before a test meal. Whey protein has been chosen as a reference protein because it has been extensively studied and its effects on blood glucose and food intake are being elucidated within our laboratory.

DETAILED DESCRIPTION:
According to the 2004 Canadian Community Health Survey, nearly two-thirds of Canadians are overweight or obese. Obesity is a major risk factor for the metabolic syndrome, which is linked to conditions such as type II diabetes. Dietary interventions that increase satiety (to promote weight loss) and maintain normal blood glucose levels are noninvasive and inexpensive compared to pharmacological strategies. Thus, it is important to identify types/sources of macronutrients that contribute to healthy body weight by increasing satiety and thereby reducing food intake. For instance, diets including pulses (legumes) have been linked with a lower risk of obesity/overweight.

Pulses are the edible seeds of legumes or pod-bearing plants including dry beans, yellow peas, lentils and chickpeas. They are inexpensive healthy foods high in protein and complex carbohydrates. Recently within our laboratory, we found that including 5 cups of pulses into the diet for 8 weeks was associated with decreased body weight, waist circumference and improved glycemic control. However, the mechanisms driving weight loss and improved glycemic control need further investigation. For instance, pulses may affect satiety, energy intake and blood glucose because of their high amounts of protein. Protein is known to be more satiating than carbohydrate and fat leading to a positive impact on long-term body weight maintenance. Protein from various animal and plant sources has also been shown to stimulate the release of satiety-related hormones like insulin, glucagon, glucagon-like peptide-1 (GLP-1), cholecystokinin (CCK), peptide tyrosine tyrosine (PYY) and ghrelin.

The investigators recently investigated the independent dosage effects of pea protein (10 and 20 g) and pea fibre (10 and 20 g) on ad libitum food intake at 30 minutes and pre- (0-30 minutes) and post-meal (50-170 minutes) blood glucose response and subjective appetite in young men. Preliminary results indicate that increasing protein amounts (10 g versus 20 g) lead to decreased pre-meal blood glucose response and reduced food intake.

Food-grade proteins are also available intact and/or hydrolyzed (partially digested through a controlled enzymatic process). Hydrolyzed proteins are more easily digested and absorbed, eliciting a faster rise in plasma amino acids compared to intact proteins and different hormonal and metabolic responses between the two forms. As for pea protein, no data are available differentiating the effects of intact and hydrolyzed forms on these blood parameters and appetite in humans. Moreover, the presence of bioactive polypeptides may be affected by protein formulation (i.e. the polypeptides may be cleaved/inactivated in hydrolyzed pea protein).

Research is needed to determine whether the effect of pea protein differs on glycemic response and appetite both pre- and post-meal based on its form (intact versus hydrolyzed) and how it compares to other well-investigated proteins. This research is preliminary and may lead to future research in other population groups, including young women and overweight individuals. These results will encourage increased consumption of pulse fractions by providing a basis for the potential use of pea protein in the development of new functional foods aimed at preventing and managing obesity along with controlling blood glucose for diabetes management. Furthermore, results will show if pea protein is a comparable alternative to whey, which would be favorable for consumers shifting away from animal-derived proteins for health and/or environmental reasons.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking
* Aged 20-30 years
* Body mass index between 20 and 24.9 kg/m2

Exclusion Criteria:

* Diabetes
* Gastrointestinal conditions
* Medication
* Lactose-intolerance or allergies to milk (standard breakfast provided)
* Breakfast skippers and those on an energy restricted diet

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Food Intake | 30 minutes

SECONDARY OUTCOMES:
Blood Glucose | 0, 15, 30, 50, 65, 80, 95, 110, 140 and 170 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, PHD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada